CLINICAL TRIAL: NCT00884221
Title: A Randomized, Open-label, Assessor-blind, Parallel Groups, Multicentre Trial Comparing the Efficacy of MENOPUR Versus Recombinant FSH in Controlled Ovarian Stimulation Following a GnRH Antagonist Protocol and Single Embryo Transfer
Brief Title: MENOPUR in Gonadotrophin-releasing Hormone (GnRH) Antagonist Cycles With Single Embryo Transfer
Acronym: MEGASET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FE999906 CS08; EudraCT Number: 2008-006775-67
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins; Glycoprotein Hormones, alpha Subunit; follitropin beta

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Highly Purified Menotrophin (Experimental)
  Interventions: Drug: Highly purified menotrophin
- Recombinant FSH (Active Comparator)
  Interventions: Drug: Recombinant FSH

INTERVENTIONS:
Drug: Highly purified menotrophin — The gonadotrophin starting dose was 150 IU daily for the first 5 days. From stimulation day 6 and onwards, dosing could be adjusted according to individual participant response. The dose adjustment could be by 75 IU per adjustment and could not be done more frequently than every 4 days. The maximum allowed gonadotrophin dose was 375 IU daily and participants could be treated with gonadotrophin for a maximum of 20 days.
  NOTE: The gonadotrophins (highly purified menotrophin and the active comparator recombinant FSH) were administered in an identical fashion.
  Other Names: HP-hMG; MENOPUR
  Arms: Highly Purified Menotrophin
Drug: Recombinant FSH — The gonadotrophin starting dose was 150 IU daily for the first 5 days. From stimulation day 6 and onwards, dosing could be adjusted according to individual participant response. The dose adjustment could be by 75 IU per adjustment and could not be done more frequently than every 4 days. The maximum allowed gonadotrophin dose was 375 IU daily and participants could be treated with gonadotrophin for a maximum of 20 days.
  NOTE: The gonadotrophins (highly purified menotrophin and the active comparator recombinant FSH) were administered in an identical fashion.
  Other Names: Follitrophin-beta; PUREGON; FOLLISTIM
  Arms: Recombinant FSH

SUMMARY:
The main purpose of this clinical research trial was to compare the ongoing pregnancy rate between two gonadotrophins for controlled ovarian stimulation (MENOPUR and recombinant follicle-stimulating hormone (FSH)), in cycles where a gonadotrophin-releasing hormone (GnRH) antagonist was used for prevention of premature luteinizing hormone (LH) surge and where a single embryo was transferred at the blastocyst stage.

DETAILED DESCRIPTION:
This was a randomized, open-label, assessor-blind, parallel groups, multicentre trial comparing the efficacy of highly purified menotrophin (MENOPUR; Ferring) and recombinant FSH (PUREGON/FOLLISTIM; MSD/Merck) in women undergoing controlled ovarian stimulation following a GnRH antagonist protocol.

The use of oral contraceptives for programming of the trial cycle was prohibited. On day 2-3 of the menstrual cycle, participants were randomized in a 1:1 fashion to treatment with either highly purified menotrophin (MENOPUR) or recombinant FSH, and stimulation was initiated.

The gonadotrophin starting dose was 150 international units (IU) daily for the first 5 days. Hereafter, the participants were seen on stimulation day 6 and subsequently at least every 2 days when a transvaginal ultrasound was made to monitor response to stimulation. From stimulation day 6 and onwards, dosing could be adjusted according to individual patient response with the purpose of achieving 8-10 oocytes at the time of oocyte retrieval. The dose adjustment could be by 75 IU per adjustment and could not be done more frequently than every 4 days. The maximum allowed gonadotrophin dose was 375 IU daily and participants could be treated with gonadotrophin for a maximum of 20 days. Coasting was prohibited.

The GnRH antagonist (ORGALUTRAN/GANIRELIX ACETATE INJECTION; MSD/Merck) was initiated on stimulation day 6 at a daily dose of 0.25 mg and continued throughout the gonadotrophin treatment period. A single injection of recombinant human chorionic gonadotrophin (hCG) 250 µg (OVITRELLE/OVIDREL; Merck Serono/EMD Serono) was administered to induce final follicular maturation as soon as 3 follicles of ≥ 17 mm were observed; i.e., the day of reaching the hCG criterion or the next day. Oocyte retrieval took place 36h (± 2h) after hCG administration. Oocytes were inseminated using partner sperm by intracytoplasmic sperm injection (ICSI) 4h (± 1h) after retrieval. Oocyte, embryo and blastocyst quality was assessed daily from oocyte retrieval till 5 days after. On day 5 after oocyte retrieval, a single blastocyst of the best quality available was transferred and all remaining blastocysts were frozen. Vaginal progesterone capsules (UTROGESTAN; Seid) 600 mg/day were provided for luteal phase support from the day after oocyte retrieval till the day of the beta human chorionic gonadotrophin (βhCG) test (13-15 days after embryo transfer); prolonged luteal phase support beyond this time point was not allowed. Clinical pregnancy was confirmed by transvaginal ultrasound 5-6 weeks after embryo transfer and ongoing pregnancy was confirmed by transvaginal ultrasound 10-11 weeks after embryo transfer. Post-trial follow-up included pregnancy outcome (e.g. live birth) and neonatal health from the fresh trial cycle. Additional post-trial activities included follow-up of frozen embryo replacement cycles initiated within 1 year after the participant's randomization date.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent Documents signed prior to screening evaluations
* In good physical and mental health
* Pre-menopausal females 21-34 years of age
* Body mass index (BMI)18-25 kg/m2
* Eligible for intracytoplasmic sperm injection (ICSI)
* Unexplained infertility or partner with mild male factor infertility
* Infertility for at least 12 months before randomization
* Regular menstrual cycles of 24-35 days, presumed to be ovulatory
* Hysterosalpingography, hysteroscopy, or transvaginal ultrasound documenting a uterus consistent with expected normal function
* Transvaginal ultrasound documenting expected normal function of the ovaries
* Early follicular phase serum levels of FSH between 1 and 12 IU/L
* Early follicular phase total antral follicle (diameter 2-10 mm) count ≥ 10 for both ovaries combined
* Willing to accept transfer of one blastocyst in the fresh cycle
* Willing to undergo frozen embryo replacement cycles with transfer of one blastocyst per cycle within the first year after randomisation

Exclusion criteria:

* Known polycystic ovarian syndrome or known endometriosis stage I-IV
* Diagnosed as "poor responder" in a previous controlled ovarian stimulation (COS) cycle
* Severe ovarian hyperstimulation syndrome (OHSS)in a previous COS cycle
* History of recurrent miscarriage
* Current or past (12 months prior to randomization) abuse of alcohol or drugs, and/or current (last month) intake of more than 14 units of alcohol per week
* Current or past smoking habit of more than 10 cigarettes per day
* Hypersensitivity to any active ingredient or excipients in the medicinal products used in the trial
* Hypersensitivity to gonadotrophin-releasing hormone (GnRH) or any other GnRH analogue
* Previous participation in the trial
* Use of any non registered investigational drugs during 3 months before randomization

Ages: 21 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 749 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (25):
- Belgium (4):
  - ERASME Hospital, Anderlecht
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
- Czechia (3):
  - IVF Institute, Pilsen
  - ISCARE IVF a.s., Prague
  - Pronatal, Prague
- Denmark (4):
  - H:S Rigshospitalet, Copenhagen
  - Amtssygehuset Herlev, Herlev
  - Sygehus Vestsjælland, Holbæk
  - H:S Hvidovre Hospital, Hvidovre
- Poland (2):
  - KRIOBANK, Bialystok
  - nOvum, Warsaw
- Spain (6):
  - IU Dexeus, Barcelona
  - GINEFIV, Madrid, Madrid
  - IVI Madrid, Madrid
  - Ginemed, Seville
  - IVI Sevilla, Seville
  - IVI Valencia, Valencia
- Sweden (3):
  - Fertilitetscentrum AB Gothenburg, Gothenburg
  - IVF-kliniken CURA, Malmo
  - RMC, Malmö, Malmo
- Turkey (Türkiye) (3):
  - Hacettepe University, Ankara
  - American Hospital, Istanbul
  - Memorial Hospital, Istanbul

REFERENCES:
- [Result] Devroey P, Pellicer A, Nyboe Andersen A, Arce JC; Menopur in GnRH Antagonist Cycles with Single Embryo Transfer Trial Group. A randomized assessor-blind trial comparing highly purified hMG and recombinant FSH in a GnRH antagonist cycle with compulsory single-blastocyst transfer. Fertil Steril. 2012 Mar;97(3):561-71. doi: 10.1016/j.fertnstert.2011.12.016. Epub 2012 Jan 13. PMID 22244781
- [Derived] Arce JC, La Marca A, Mirner Klein B, Nyboe Andersen A, Fleming R. Antimullerian hormone in gonadotropin releasing-hormone antagonist cycles: prediction of ovarian response and cumulative treatment outcome in good-prognosis patients. Fertil Steril. 2013 May;99(6):1644-53. doi: 10.1016/j.fertnstert.2012.12.048. Epub 2013 Feb 5. PMID 23394782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited among the patients attending the clinics included in the trial.
Pre-assignment Details: 810 participants were screened and 754 were randomised. 749 participants were exposed to highly purified menotrophin or recombinant FSH
Groups:
- Highly Purified Menotrophin; Recombinant FSH: The gonadotrophin starting dose was 150 IU daily for the first 5 days. Hereafter, the subjects were seen on stimulation day 6 and subsequently at least every 2 days when a transvaginal ultrasound was made to monitor response to stimulation. From stimulation day 6 and onwards, dosing could be adjusted according to individual patient response with the purpose of achieving 8-10 oocytes at the time of oocyte retrieval. The dose adjustment could be by 75 IU per adjustment and could not be done more frequently than every 4 days. The maximum allowed gonadotrophin dose was 375 IU daily and subjects could be treated with gonadotrophin for a maximum of 20 days. Coasting was prohibited.
Period: Overall Study
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Started | 374 | 375
Completed | 340 | 343
Not Completed | 34 | 32
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 6 | 3
Not completed — Protocol Violation | 16 | 13
Not completed — Cancellation of Cycle and Other Reason | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Highly Purified Menotrophin; Recombinant FSH: The gonadotrophin starting dose was 150 IU daily for the first 5 days. From stimulation day 6 and onwards, the dosing could be adjusted according to individual patient response with the purpose of achieving 8-10 oocytes at the time of oocyte retrieval. The dose adjustment could be by 75 IU per adjustment and could not be done more frequently than every 4 days. The maximum allowed gonadotrophin dose was 375 IU daily and subjects could be treated with gonadotrophin for a maximum of 20 days.
- Total: Total of all reporting groups
Arm/Group | Highly Purified Menotrophin | Recombinant FSH | Total
Number analyzed (Participants) | 374 | 375 | 749
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 374 | 375 | 749
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.8 (2.75) | 30.4 (2.62) | 30.6 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 375 | 749
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 20 | 20 | 40
  Czech Republic | 30 | 27 | 57
  Denmark | 33 | 33 | 66
  Poland | 72 | 71 | 143
  Spain | 179 | 178 | 357
  Sweden | 14 | 19 | 33
  Turkey | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy After One Fresh Embryo Replacement Cycle, Intention-to-treat (ITT) Analysis Set
Description: Transvaginal ultrasound showing at least one intrauterine viable fetus 10-11 weeks after embryo transfer at the blastocyst stage
Time Frame: 10-11 weeks after embryo transfer at the blastocyst stage
Population: The intention-to-treat (ITT) analysis set was defined as all randomized and exposed participants. Participants were analyzed according to actual treatment.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Groups:
- Highly Purified Menotrophin; Recombinant FSH: The gonadotrophin starting dose was 150 IU daily for the first 5 days. From stimulation day 6 and onwards, the dosing could be adjusted according to individual participant response with the purpose of achieving 8-10 oocytes at the time of oocyte retrieval. The dose adjustment could be by 75 IU per adjustment and could not be done more frequently than every 4 days. The maximum allowed gonadotrophin dose was 375 IU daily and participants could be treated with gonadotrophin for a maximum of 20 days.
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Percentage of participants | 29 (2.3) [-4.2 to 8.6] | 27 (2.3)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; The non-inferiority hypothesis to be tested for the primary endpoint was: H0: π MENOPUR - π recombinant FSH ≤ -10.0% against the alternative H1: π MENOPUR - π recombinant FSH > -10.0%, where π MENOPUR and π recombinant FSH denote the ongoing pregnancy rate after treatment with MENOPUR and recombinant FSH, respectively, in a single fresh treatment cycle following a GnRH antagonist protocol; Test type: Non-Inferiority or Equivalence — The null hypothesis (H0) was tested against the alternative by constructing a two-sided 95% confidence interval for the difference in ongoing pregnancy rates. If the lower-limit of the 95% confidence interval was greater than the non-inferiority limit (-10.0%), the null hypothesis was rejected and it would be claimed that highly purified menotrophin was non-inferior to recombinant FSH with respect to ongoing pregnancy rate in a single fresh treatment cycle following a GnRH antagonist protocol; p = 0.499, Sign test — Since there was only one primary endpoint, no adjustment for multiplicity was needed for the primary analysis; A two-sided 95% confidence interval for the difference in ongoing pregnancy rates was made. The CI was based on a normal approximation; Difference in pregnancy rates, ITT = 2.2, 95% CI 2-sided [-4.2 to 8.6] — Difference tested: highly purified menotrophin-recombinant FSH, ITT analysis set

2. Secondary Outcome: Endocrine Profile (Estradiol), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: On the last day of stimulation, blood was drawn at least 8 hours after the previous injection of gonadotrophin and GnRH antagonist
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
pmol/L | 8797 (6030) [4993 to 10136] | 7022 (4945) [4023 to 8234]
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Estradiol; Test type: Superiority or Other; p < 0.001, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

3. Secondary Outcome: Endocrine Profile (FSH), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
IU/L | 15.7 (4.1) | 12.6 (3.7)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; FSH; Test type: Superiority or Other; p < 0.001, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

4. Secondary Outcome: Endocrine Profile (Free Androgen Index), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn. Free androgen index = (testosterone (nmol/L)/ sex hormone binding globulin (nmol/L))*100
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Percentage of participants | 2.8 (2.0) | 2.5 (2.2)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Free Androgen Index; Test type: Superiority or Other; p < 0.001, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

5. Secondary Outcome: Endocrine Profile (Luteinizing Hormone), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
IU/L | 2.8 (2.8) | 2.1 (1.6)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Luteinizing hormone; Test type: Superiority or Other; p < 0.001, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

6. Secondary Outcome: Endocrine Profile (Progesterone), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
nmol/L | 3.1 (3.4) | 3.1 (3.3)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Progesterone; Test type: Superiority or Other; p = 0.630, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

7. Primary Outcome: Ongoing Pregnancy After One Fresh Embryo Replacement Cycle, Per-protocol (PP) Analysis Set
Description: as for outcome 1
Time Frame: 10-11 weeks after embryo transfer at the blastocyst stage
Population: The per-protocol (PP) analysis set was defined as all randomized and exposed participants except those excluded as a result of major protocol deviations, such as significant non-compliance or other serious unforeseen deviations deemed to invalidate the data and affect the conclusions of the trial.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 343 | 333
Percentage of participants | 30 (2.5) | 27 (2.4)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.387, Sign test — Since there was only one primary endpoint, no adjustment for multiplicity was needed for the primary analysis; [statistical method as in outcome 1, analysis 1]; Difference in pregnancy rates, PP = 3.0, 95% CI 2-sided [-3.8 to 9.8] — Difference tested: highly purified menotrophin - recombinant FSH, PP

8. Secondary Outcome: Endocrine Profile (Prolactin), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
pmol/L | 1544 (770) | 1410 (689)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Prolactin; Test type: Superiority or Other; p = 0.047, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

9. Secondary Outcome: Endocrine Profile (Sex Hormone Binding Globulin), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
nmol/L | 111 (51) | 107 (48)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Sex hormone binding globulin; Test type: Superiority or Other; p = 0.009, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

10. Secondary Outcome: Endocrine Profile (Testosterone), Intention-to-treat (ITT) Analysis Set
Description: Blood samples for analysis of circulating concentrations of endocrine parameters were drawn
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
nmol/L | 2.5 (1.2) | 2.1 (1.0)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Testosterone; Test type: Superiority or Other; p < 0.001, Regression, Linear; Tests for treatment differences were based on log-transformed values and adjusted for baseline values

11. Secondary Outcome: Number of Follicles of >= 12mm, 12-14 mm, 15-16 mm and >= 17 mm in Each Participant, Intention-to-treat (ITT) Analysis Set
Description: During the controlled ovarian stimulation, transvaginal ultrasound was performed to count the number of follicles and measure the size of the follicles.
Time Frame: Last stimulation day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Follicles per participant
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Follicles per participant
  >= 12 mm | 10.9 (4.7) | 11.8 (4.9)
  12-14 mm | 3.3 (2.6) | 3.8 (2.9)
  15-16 mm | 2.7 (2.2) | 2.7 (2.3)
  >=17 mm | 4.9 (2.2) | 5.2 (2.4)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatment groups of the average number of follicles >= 12 mm on the last stimulation day; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatment groups of the average number of follicles 12-14 mm on the last stimulation day; Test type: Superiority or Other; p = 0.024, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatment groups of the average number of follicles 15-16 mm on the last stimulation day; Test type: Superiority or Other; p = 0.728, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatment groups of the average number of follicles >=17 mm on the last stimulation day; Test type: Superiority or Other; p = 0.285, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Number of Oocytes Retrieved in Each Participant, Intention-to-treat (ITT) Analysis Set
Description: Oocyte retrieval took place 36h (± 2h) after hCG administration. At oocyte retrieval, the number of oocytes retrieved was recorded.
Time Frame: 36 h after hCG
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Oocytes per participant
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Oocytes per participant | 9.1 (5.2) | 10.7 (5.8)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Treatments were compared using the Wilcoxon test for the average number of oocytes retrieved; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Only participants who underwent the oocyte retrieval procedure were included in the analysis

13. Secondary Outcome: Fertilization, Intention-to-treat (ITT) Analysis Set
Description: Fertilized oocytes with 2 pronuclei were regarded as correctly fertilized. Fertilization was estimated as (Number of oocytes with 2 pronuclei / number of metaphase II oocytes)*100
Time Frame: 1 day after oocyte retrieval (19 h post-insemination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of metaphase II oocytes
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Percentage of metaphase II oocytes | 75 (23) | 76 (22)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Test type: Superiority or Other; p = 0.969, Wilcoxon (Mann-Whitney); Only participants who had oocytes retrieved were included in the analysis

14. Secondary Outcome: Blastocyst Quality, Intention-to-treat (ITT) Analysis Set
Description: Blastocyst quality on day 5 was based on the blastocyst expansion and hatching status, inner cell mass grading and trophectoderm grading.
  Excellent-quality blastocysts were defined as those with blastocyst expansion and hatching status 4, 5 or 6, inner cell mass grading A, and trophectoderm grading A or B. Good-quality blastocysts were defined as those with blastocyst expansion and hatching status 3, 4, 5 or 6, inner cell mass grading A or B, and trophectoderm grading A or B.
Time Frame: 5 days after oocyte retrieval (120h post-insemination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of blastocysts
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Number of blastocysts
  Blastocyst 1 / 2 pn | 7 (17) | 7 (16)
  Blastocyst 2 / 2pn | 7 (15) | 5 (11)
  Blastocyst 3 / 2pn | 10 (16) | 10 (15)
  Blastocyst 4 / 2pn | 18 (22) | 20 (26)
  Blastocyst 5 / 2pn | 7 (16) | 6 (13)
  Blastocyst 6 / 2pn | 0 (0) | 0 (0)
  Blastocyst 4AA/ 2pn | 5 (13) | 5 (14)
  Blastocyst 5AA / 2pn | 2 (7) | 2 (7)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status 1 / 2pn; Test type: Superiority or Other; p = 0.406, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status 2 / 2pn; Test type: Superiority or Other; p = 0.232, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status 3 / 2pn; Test type: Superiority or Other; p = 0.412, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status 4 / 2pn; Test type: Superiority or Other; p = 0.438, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status 5 / 2pn; Test type: Superiority or Other; p = 0.390, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status, inner cell mass grading and trophectoderm grading 4AA / 2pn; Test type: Superiority or Other; p = 0.958, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Comparison between treatments groups of percentage of blastocysts with expansion and hatching status, inner cell mass grading and trophectoderm grading 5AA / 2pn; Test type: Superiority or Other; p = 0.954, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Live Birth for a Single Stimulation Cycle With Single Blastocyst Transfer From Fresh Embryo Replacement Cycle, Intention-to-treat (ITT) Analysis Set
Time Frame: Post-trial information
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Percentage of participants | 28 (2.3) | 26 (2.3)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Test type: Superiority or Other; p = 0.398, Wilcoxon (Mann-Whitney); A two-sided 95% confidence interval for the difference in live birth rates was made. The CI was based on a normal approximation; Comparison of distributions = 0.398, 95% CI 2-sided [-3.6 to 9.1] — Estimated value is difference between highly purified menotrophin and recombinant FSH, ITT analysis set

16. Secondary Outcome: Cumulative Live Birth for a Single Stimulation Cycle With Single Blastocyst Transfer From Fresh and 1 Year Frozen Embryo Replacement Cycles, Intention-to-treat (ITT) Analysis Set
Time Frame: Post-trial information
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Number analyzed (Participants) | 374 | 375
Percentage of participants | 40 (2.5) | 38 (2.5)
Statistical Analysis 1: Comparison: Highly Purified Menotrophin vs Recombinant FSH; Test type: Superiority or Other; p = 0.686, Wilcoxon (Mann-Whitney); A two-sided 95% confidence interval for the difference in cumulative live birth rates was made. The CI was based on a normal approximation; Comparison of distributions = 1.8, 95% CI 2-sided [-5.6 to 9.2] — Estimated value is difference between highly purified menotrophin and recombinant FSH, ITT analysis set

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signed informed consent until the end-of-trial visit.
Description: Adverse events were evaluated at each visit.
Arm/Group | Highly Purified Menotrophin | Recombinant FSH
Serious Adverse Events (participants affected / at risk) | 5/374 | 7/375
Other Adverse Events (participants affected / at risk) | 66/374 | 47/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Highly Purified Menotrophin (N=374) | Recombinant FSH (N=375)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Highly Purified Menotrophin (N=374) | Recombinant FSH (N=375)
Nausea (Gastrointestinal disorders) | 18 (19) | 15 (16)
Headache (Nervous system disorders) | 25 (30) | 19 (23)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 27 (27) | 19 (19)
Pelvic pain (Reproductive system and breast disorders) | 18 (23) | 16 (20)
Vaginal haemorrhage (Reproductive system and breast disorders) | 21 (25) | 10 (13) — Episodes of vaginal haemorrhage mainly covered episodes of vaginal bleeding during pregnancy not associated with pregnancy loss; no episodes during ovarian stimulation with highly purified menotrophin or recombinant FSH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the principle investigator (PI) is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.